CLINICAL TRIAL: NCT05237141
Title: Etonogestrel Implant as Emergency Contraception: A Pilot Pharmacodynamic Study
Brief Title: Etonogestrel Implant as Emergency Contraception
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-5026
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main cohort (Experimental): Insertion of etonogestrel contraceptive implant prior to LH surge
  Interventions: Drug: Etonogestrel implant

INTERVENTIONS:
Drug: Etonogestrel implant — Implant insertion in second menstrual cycle prior to ovulation

SUMMARY:
The investigators propose a single site, single arm, open label mechanism of action pharmacodynamic pilot study of etonogestrel implant insertion prior to an luteinizing hormone (LH) surge. The investigators will evaluate ovulation rates via serum levels of reproductive hormones and transvaginal ultrasound findings following placement of an etonogestrel implant once the dominant follicle reaches a size of 15mm or greater, but prior to an LH surge, in persons with prior documented regular cycles and confirmed ovulation. The researchers' hypothesis is that ovulation will be inhibited if the etonogestrel implant is placed prior to an LH surge.

Based on data from the Food and Drug Administration label for Nexplanon, etonogestrel rises to levels associated with ovulation suppression within 8 hours of placement. Given this rapid increase, it is therefore plausible to assume that ovulation can be inhibited by the implant if placed prior to an LH surge. This study is novel as there have been no published studies evaluating an etonogestrel implant for this indication.

The contribution of this proposed research to the literature is significant because current recommendations from the Center for Disease Control (CDC) regarding timing of etonogestrel implant placement are stringent and not patient-centered. Any day insertion of the etonogestrel implant is supported by retrospective data and this pharmacodynamic data would further support the literature for any day insertion without the need for additional emergency contraception. If results support the investigators' hypothesis, it could increase access to contraception and decrease duplicative therapy.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than or equal to 28kg/m2
* Intact uterus with at least one ovary
* Regular menstrual cycles that occur every 21-35 days
* If patient is postpartum or post-second trimester abortion, 3 menses (2 cycles) must have occurred prior to enrollment
* If patient had a first trimester abortion or pregnancy loss, she must have one spontaneous menses prior to enrollment
* Desires insertion of an etonogestrel contraceptive implant for contraception
* Not currently pregnant or trying to become pregnant
* Willing to abstain from medications and supplements known to induce/inhibit CYP3A4 during the study

Exclusion Criteria:

* Have a known hypersensitivity or contraindications to etonogestrel.
* Medical conditions that affect liver function (e.g., hepatitis, cirrhosis; assessed via participant self-report)
* Known or suspected current alcohol dependence syndrome or any illicit drug use that may affect the metabolism of the etonogestrel.
* Uncontrolled thyroid disorder.
* Use of long-acting injectable hormonal contraceptive within the past 9 months
* Current use of hormonal oral, patch, intravaginal, or intrauterine contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serum progesterone | 7 days
  Serial measurements of serum progesterone will be conducted after insertion of the etonogestrel implant to assess for evidence of potential ovulation (>3ng/mL)
Ovarian follicle size | 7 days
  Serial transvaginal ultrasound measurements of the leading or dominant follicle will be conducted after insertion of the etonogestrel implant. Ovulation will be defined by follicle rupture with complete disappearance or at least a 50% reduction in the mean size of the leading follicle.

SECONDARY OUTCOMES:
Luteinizing hormone | 7 days
  Serial measurements of serum luteinizing hormone will be conducted after insertion of the etonogestrel implant. These LH concentrations will be used to support the primary outcomes in assessing ovulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Will share summary data if requested